CLINICAL TRIAL: NCT00335712
Title: Phase II Study of ONO-5129 in Patients With Type 2 Diabetes Mellitus
Brief Title: Pilot Study of ONO-5129 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5129-03
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: ONO-5129; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: ONO-5129

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of ONO-5129 in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting Blood Glucose 126-250mg/dL
2. HbA1c 6.5-11%

Exclusion Criteria:

1. Previous treatment with antidiabetic agents equal to or less than 2-3 months prior to randomization
2. History of myocardial infarction, coronary artery surgery
3. Other eligibility criteria as specified in the study protocol

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Fasting Blood Glucose at week 8

SECONDARY OUTCOMES:
Other glycemic control parameters (e.g., HbA1c, glycoalbumin)

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (2):
- Japan (2):
  - Kanto Region, Kanto
  - Kyusyu Region, Kyusyu